CLINICAL TRIAL: NCT06724393
Title: Demonstrating the Effects of Blood Flow Restriction During Resistance Training on Functionality, Strength and Oxygen Capacity in Older Adults
Brief Title: Blood Flow Restriction and Functionality in Older Adults
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Concordia University, Montreal (Other)
Responsible Party: Principal Investigator, Andreas Bergdahl, Associate Professor, Concordia University, Montreal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 30018588
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Older Adults (65 Years and Older); Older Adults At Risk of Falling; Blood Flow Restriction (BFR) Training Effects; Blood Flow Restriction and Low-Intensity Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): This group with undergo online low-intensity resistance training twice per week
  Interventions: Other: Blood flow restrictions in combination with low-intensity resistance training
- Blood flow restriction (Experimental): This group with undergo online low-intensity resistance training with blood flow restriction twice per week
  Interventions: Other: Blood flow restrictions in combination with low-intensity resistance training

INTERVENTIONS:
Other: Blood flow restrictions in combination with low-intensity resistance training — Blood flow restrictions in combination with low-intensity resistance training to test if an online intervention (telehealth) can improve functional capacity and balance in older adults

SUMMARY:
Resistance training is beneficial for stimulating muscle and bone growth and is uniquely important for older adults to avoid frailty and to maintain bone density. Seniors tend to be anxious to use a large resistance or try heavier weights as it is not common for them to exercise this way. Therefore, blood flow restriction is a fantastic way to increase intensity while keeping the resistance low. Wearing blood flow restriction straps allows the muscles to adapt to working at a lower oxygen pressure, therefore, mimicking a higher intensity. Additionally, as we age, oxygen consumption decreases, commonly due to loss of lean body mass and a reduced maximum heart rate. However, resistance training can counteract these declines by reducing the resting heart rate and improving cardiac output, therefore, bettering oxygen consumption.

The study will consist of 10 weeks of resistance exercises performed twice per week. The classes will be open to seniors of 60 years of age or older. The classes will be held on zoom- allowing for easy access, no travel and an opportunity for seniors to be active in their own home. The exercises will consist of general resistance training movements focusing all the major muscle groups. One group of seniors will wear blood flow restriction bands on both legs at the upper thigh and a control group which will complete the same exercise classes with no restriction.

Before, at midpoint and after the 10 weeks, the participants will perform strength tests using the BIODEX and three functional tests focusing on the lower extremity. There will be a practice trial for all the functional tests where results are not recorded. Once the practice is completed, the participants will have one trial of each test. The BIODEX is a dynamometer that allows testing in many different settings including rehabilitation. During the functional tests, the participants will be asked to wear a VO2 non-invasive mask (VO2 Master) to measure their oxygen consumption. The functional tests will include:

* Sit to stand: rise from a chair as many times as possible without using hands or arm rests to help.
* Timed up a go: Rise from a chair and walk 8ft as fast as possible without running and return to sit on the chair.
* Sitting-rising test: lowering to the floor and coming back up without using hands, knees or arms.

Thus, the purpose of this study is three-fold: 1) To assess the effects of the 10-week online exercise intervention on strength and functionality 2) To assess the effects of the 10-week intervention on oxygen consumption using a VO2 non-invasive mask and 3) To assess if the addition of blood flow restriction over a 10-week intervention increases the improvements in strength and oxygen consumption compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be both male and female, aged 60 years or older. They must be willing to participate in two exercise sessions per week for 10 weeks held online. Participants must also be able to visit Loyola campus for pre-, mid- and post-intervention testing.

Exclusion Criteria:

* Exclusion criteria include chronic disease (with the exclusion of hypertension), use of steroidal drugs, blood clot or varicose veins, part-take in excessive physical activity (over 3-4 hours a week of moderate to high intensity training) and have scheduled vacation or absence in the ten-week period. The reason behind excluding seniors who part-take in excessive physical activity is because the classes will be low intensity. Due to the fact that participants will be healthy older adults without chronic conditions, a medical form from a physician will not be necessary.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Functional capacity | From enrollment to the end of intervention at 10 weeks

SECONDARY OUTCOMES:
Balance and posture | From enrollment to the end of intervention at 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Concordia University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Presta D, Bergdahl A. 5 weeks of online resistance training with blood flow restriction increases sit-to-stand oxygen consumption in healthy older adults. Can J Physiol Pharmacol. 2026 Jan 19. doi: 10.1139/cjpp-2025-0270. Online ahead of print. PMID 41565628